CLINICAL TRIAL: NCT03656211
Title: Fertility After Diagnosis and Management of Acquired Uterine Arteriovenous Malformation
Acronym: MAVUFERT
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3026; 2017-A01760-53 (Other: Id-RCB)
Record Dates: First submitted 2018-08-29; First posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Arteriovenous Malformations
Keywords: Uterine AVM
MeSH Terms: conditions — Arteriovenous Malformations | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with UAVM: All patients who have been diagnosed with UAVM (symptomatic or non-symptomatic) between January 1, 2000 and March 30, 2017, and confirmed by an imaging examination.
  Telephone interview
  Interventions: Other: Telephone interview

INTERVENTIONS:
Other: Telephone interview — Patients are contacted by telephone to know the history of the disease since the diagnosis of UAVM and the impact of management on fertility.
  All medical data related to the care and necessary for the study are collected from the medical file the participation of the patients is limited to a telephone interview.

SUMMARY:
Uterine arteriovenous malformations (UAVM) are short circuits between systemic arterial and venous networks within the uterus. They are congenital or acquired (in the course of an endo-uterine gesture such as curettage or interventions such as caesareans or myomectomies).

They can be manifested by severe metrorrhagia that can go as far as to put the patient's vital prognosis at risk.

There are no recommendations for the management of UAVM since this pathology is rare and therefore series are performed with few cases. If some of these UAVM disappear spontaneously after a therapeutic abstention, when the clinical context allows it, in case of symptomatic UAVM, a selective embolization with arteriography is often carried out to postpone the hysterectomy of hemostasis.

There are also more marginal management options such as Gonadotropin-Releasing Hormone agonists, methotrexate or curettage that are decided on a case by case basis depending on the symptoms and protocols of each medical team.

Regarding subsequent fertility and pregnancy outcomes after conservative treatment, the number of studies is even lower.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Diagnosis of UAVM, symptomatic or not, between January 1st, 2000 and March 30th, 2017 confirmed by imagery performed at the Rennes University Hospital
* Not against her participation in research

Exclusion Criteria:

* Minor patient at the time of diagnosis
* congenital UAVM
* Uterine malformation
* Patient under legal protection (guardianship, curatorship, safeguard of justice).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients having a diagnosis of UAVM posed between January 1st, 2000 and March 30th, 2017, and confirmed by an imaging examination carried out at the Rennes University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of fertility | At the time of inclusion
  The telephone interview seeks to assess fertility for all patients diagnosed with symptomatic or non-symptomatic UAVM regardless of initial management.

SECONDARY OUTCOMES:
Pregnancy outcomes after UAVM | At the time of inclusion
  The telephone interview allows to evaluate pregnancy outcomes after diagnosis of UAVM regardless of initial management, in terms of live birth (full term or preterm birth), stillbirth, spontaneous abortion, and induced abortion.
Term of delivery after UAVM | At the time of inclusion
  The telephone interview allows to evaluate the term of delivery after diagnosis of UAVM regardless of initial management
Side effects of treatments for UAVM | At the time of inclusion
  The telephone interview allows to inventory the side effects of treatments
Complications of treatments for UAVM | At the time of inclusion
  The telephone interview allows to evaluate the complications of treatments

CONTACTS AND LOCATIONS:
Overall Officials: Krystel NYANGOH-TIMOH, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided